CLINICAL TRIAL: NCT03729427
Title: Erector Spinae Plane Block for Rib Cartilage Graft Reconstruction Surgery
Brief Title: Rib Microtia and the Erector Spinae Plane (ESP) Block
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled in the study due to numerous transitions of research staff and support since 2018.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor-Med Ctr Line, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 45160
Record Dates: First submitted 2018-10-29; First posted 2018-11-02 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Microtia, Congenital; Microtia; Anesthesia, Local; Anesthesia
Keywords: Erector Spinae Plane; Erector Spiane Plane Block; Rib Cartilage
MeSH Terms: conditions — Congenital Microtia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): ESP Block
  Interventions: Procedure: Erector Spinae Plane Block
- Control Arm (No Intervention): Standard of Care

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Erector Spinae Plane block for patents undergoing rib cartilage grafting surgeries
  Arms: Treatment Arm

SUMMARY:
The erector spinae plane block is a novel regional anesthetic technique that allows for analgesia of the thorax and abdomen with a peripheral nerve block. This study is being performed to assess the effectiveness of this technique in reducing post-operative pain scores and opiate requirements in pediatric and adult patients undergoing rib cartilage grafting surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2-17
* Able to consent (if greater than 7 years) and have parental consent
* Pediatric patients undergoing rib cartilage resection surgeries

Exclusion Criteria:

* Participants who do not consent or have parental consent
* Patients who are clinically unstable or requires urgent/emergent intervention

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Opiate Intake in Morphine Equivalents in Both Control and Treatment Group | Duration of procedure and postoperative recovery (throughout study completion, typically 4-5 days)
Evaluating Pain Scores Using 0-10 Numeric Pain Scale (0=No Pain, 10=Worst Pain) | Duration of Study (Typically 4-5 days)
  Scale will be used to asses pain initially prior to the procedure and postoperatively approximately every 6 hours.
Evaluating Pain Scores Using Wong-Baker FACES Pain Rating Scale | Duration of Study (Typically 4-5 days)
  Scale will be used to asses pain initially prior to the procedure and postoperatively approximately every 6 hours.
Evaluating Pain Scores Using Faces, Legs, Activity, Cry, and Consolability (FLACC) Scale | Duration of Study (Typically 4-5 days)
  Scale will be used to asses pain initially prior to the procedure and postoperatively approximately every 6 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Erector spinae plane (ESP) block in the management of post thoracotomy pain syndrome: A case series. Scand J Pain. 2017 Oct;17:325-329. doi: 10.1016/j.sjpain.2017.08.013. Epub 2017 Sep 12. PMID 28919152
- [Background] Luftig J, Mantuani D, Herring AA, Dixon B, Clattenburg E, Nagdev A. Successful emergency pain control for posterior rib fractures with ultrasound-guided erector spinae plane block. Am J Emerg Med. 2018 Aug;36(8):1391-1396. doi: 10.1016/j.ajem.2017.12.060. Epub 2017 Dec 28. PMID 29301653
- [Background] Hamilton DL, Manickam B. Erector spinae plane block for pain relief in rib fractures. Br J Anaesth. 2017 Mar 1;118(3):474-475. doi: 10.1093/bja/aex013. No abstract available. PMID 28203765